CLINICAL TRIAL: NCT05873400
Title: Effect of Renin Angiotensin Aldosterone System Genetic Polymorphism on the Pharmacological Effect of Mineralocorticoid Receptor Antagonists in Patients With Myocardial Infarction
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Isel Alansary, Academic Researcher, Misr International University
Other Study IDs: 95
Record Dates: First submitted 2023-05-16; First posted 2023-05-24 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Myocardial Infarction
Keywords: Aldosterone Antagonist; Myocardial Infarction; Cardiac remodeling; Gene polymorphism; Remodeling Marker; Stress Marker
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- 1: Myocardial Infarction patients who responded to aldosterone antagonist and didn't develope heart failure
- 2: Myocardial Infarction patients who didn't respond to aldosterone antagonist and developed heart failure
- 3: Control group who didn't receive aldosterone antagonist

SUMMARY:
Early treatment of Myocardial Infarction patients with mineralocorticoid receptor antagonist with help reduces the incidence of cardiac remodeling and development into heart failure. Also studying aldosterone synthase (CYP11B2) and mineralocorticoid receptor (NR3C2) gene polymorphisms in Egyptian Myocardial Infarction patients will help tailor medication therapy and optimize therapeutic effects with the least adverse effects.

ELIGIBILITY:
Inclusion Criteria:

* ST- segment elevation patients.
* Patients who are candidate for add-on treatment with Mineralocorticoid receptor antagonists (MRAs) to improve cardiac remodeling.
* Age of 18 years to 80 years.
* Written informed consent of the subject to participate in the study.

Exclusion Criteria:

* Contraindications to Mineralocorticoid receptor antagonists (MRA) including: serum potassium >5.5 mEq/L at initiation; CrCl ≤30 mL/minute; concomitant use of strong CYP3A4 inhibitors; concomitant use with potassium supplements or potassium-sparing diuretics.
* Mild-to-severe valvular stenosis or severe (grade III/IV) valvular regurgitation
* Pregnant or nursing women.
* Non cardiac disorders associated with increased growth factor (e.g., HIV, Alzheimer, Crohn's disease, Cancer, glomerulonephritis, glomerulosclerosis, diabetic nephropathy, muscle atrophy, fibrotic conditions and burns).
* Patients with chronic heart failure with reduced ejection fraction (LVEF <40%).

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Myocardial Infarction patients taking Aldosterone antagonist
Sampling Method: Probability Sample
Enrollment: 102 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Genetic polymorphism | 3 months
  To investigate impact of genetic polymorphism in aldosterone synthase (CYP11B2), mineralocorticoid receptor (NR3C2) on pharmacological effect of MRAs in patients with STEMI through measurement of biochemical serum markers such as serum aldosterone, oxidative stress markers and cardiac remodeling markers.

SECONDARY OUTCOMES:
Gene Interaction | 3 months
  To investigate the potential interaction between these target gene polymorphisms and the overall patients' clinical outcome in response to treatment with Mineralocorticoid receptor antagonists (MRAs).
Gene incidence | 3 months
  To detect the incidence of aldosterone synthase (CYP11B2) and mineralocorticoid receptor (NR3C2) gene polymorphisms in Egyptian patients with ST- segment elevation (STEMI).

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No